CLINICAL TRIAL: NCT03482830
Title: Perioperative Metabolic and Hormonal Aspects in Major Emergency Surgery
Acronym: PHASE
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PHASE
Record Dates: First submitted 2018-02-13; First posted 2018-03-29 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Surgery--Complications; Acute Illness; Gastrointestinal Disease; Stress
Keywords: Inflammation; Insulin-glucose homeostasis; Hypothalamic-pituitary-adrenal axis; Endothelial function and damage; Thyroid hormones
MeSH Terms: conditions — Gastrointestinal Diseases; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Major emergency gastrointestinal surgery — * Open, laparoscopic, or laparoscopically-assisted procedures
  * Procedures involving the stomach, small or large bowel, or rectum for conditions such as perforation, ischaemia, abdominal abscess, bleeding or obstruction

SUMMARY:
Emergency laparotomies, which most often is performed due to high risk disease (bowel obstruction, ischemia, perforation, etc.), make up 11 % of surgical procedures in emergency surgical departments, however, give rise to 80 % of all postoperative complications. The 30-day mortality rates in relation to these emergent procedures have been reported between 14-30 %, with even higher numbers for frail and older patients. The specific reasons for these outcomes are not yet known, however, a combination of preexisting comorbidities, acute illness, sepsis, and the surgical stress response that arise during- and after the surgical procedure due to the activation of the immunological and humoral system, is most likely to blame. The complex endocrinological response and consequences of this response to emergency surgery are sparsely reported in the literature.

The aim of this PHASE project is to evaluate and describe the temporal endocrine, endothelial and immunological changes after major emergency abdominal surgery, and to associate these changes with clinical postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Surgery within 72 hours of an acute admission to the Department of Surgery or an acute reoperation.
* Major gastrointestinal surgery on the gastrointestinal tract (see intervention definition)

Exclusion Criteria:

* Not capable of giving informed consent after oral and written information
* Previously included in the trial
* Elective laparoscopy
* Diagnostic laparotomy/laparoscopy where no subsequent procedure is performed (NB, if no procedure is performed because of inoperable pathology, then include)
* Appendectomy +/- drainage or Cholecystectomy +/- drainage of localized collection unless the procedure is incidental to a non-elective procedure on the GI tract
* Non-elective hernia repair without bowel resection.
* Minor abdominal wound dehiscence unless this causes bowel complications requiring resection
* Ruptured ectopic pregnancy, or pelvic abscesses due to pelvic inflammatory disease
* Laparotomy/laparoscopy for pathology caused by blunt or penetrating trauma, esophageal pathology, pathology of the spleen, renal tract, kidneys, liver, gall bladder and biliary tree, pancreas or urinary tract

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 18 years old undergoing acute major gastrointestinal surgery within 72 hours of their admission to the Department of Surgery or an acute reoperation.
  Major gastrointestinal surgery are defined as procedures involving the stomach, small or large bowel, or rectum for conditions such as perforation, ischaemia, abdominal abscess, bleeding or obstruction.
  Patients will be consecutively screened for inclusion.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Changes of immunological biomarkers | Change from preoperative levels at postoperative day 5
  Assessment of:
  * plasma inflammatory interleukines incl. IL-1-alfa, IL-1beta, IL-6, IL-10
  * plasma TNF-alfa
  * plasma TGF-beta
Number of patients with stress induced hyperglycemia | Postoperative day 5
  Assessment of:
  * Blood glucose, plasma c-peptide, HbA1C
  * plasma Glucagon-like peptide 1 (GLP-1)
Changes of plasma thyroid hormones | Change from preoperative levels at postoperative day 5
  Assessment of:
  * Thyropin-releasing hormone (TRH)
  * Thyroid-stimulating hormone (TSH)
  * Thyroid hormones (fT3, fT4, rT3)
Changes of the central endocrine stress response | Change from preoperative levels at postoperative day 5
  Assessment of plasma corticotropin releasing hormone (CRH)
Changes of sE-selectin | Change from preoperative levels at postoperative day 5
  Assessment of plasma sE-selectine
  * sE-selectin
  * syndecan-1
  * thrombomodulin
  * sVE-cadherin
Changes of the endothelial function | Change from postoperative day 1 at postoperative day 5
  Assessed with the non-invasive EndoPAT and expressed as the reactive hyperemia index
Changes of the periferal endocrine stress response | Change from preoperative levels at postoperative day 5
  Assessment of plasma adrenocorticotropic hormone (ACTH)
Changes of cortisol | Change from preoperative levels at postoperative day 5
  Assessment of plasma cortisol (free and bound)
Changes of neuropeptides | Change from preoperative levels at postoperative day 5
  Assessment of plasma neuropeptides
Changes of syndecan-1 | Change from preoperative levels at postoperative day 5
  Assessment of plasma syndecan-1
Changes of thrombomodulin | Change from preoperative levels at postoperative day 5
  Assessment of plasma thrombomodulin
Changes of sVE-cadherin | Change from preoperative levels at postoperative day 5
  Assessment of plasma sVE-cadherin

SECONDARY OUTCOMES:
Number of patients with major adverse cardiovascular events | 365 days after surgery
  Defined as:
  * Cardiovascular death
  * Myocardial injury within postoperative day 4 (definition: peak plasma cardiac troponin-I ≥ 45ng/L (99th percentile URL, 10% CV at 40ng/L))
  * Acute coronary syndrome (unstable angina pectoris, NSTEMI, STEMI)
  * Congestive heart failure
  * Stroke
  * Nonfatal cardiac arrest
  * New clinically important cardiac arrhythmia
  * Coronary revascularization procedure (PCI or CABG)
  * Sudden unexpected death
Number of patients with postoperative non-cardiovascular complications | 365 days after surgery
  Defined as:
  * Non-cardiovascular death with other defined reason for death
  * Sepsis (sepsis - severe sepsis - septic shock)
  * Pneumonia
  * Respiratory failure
  * Surgical complications (Clavien-Dindo stage 3)
  * Any non-cardiovascular life-threatening complication (Clavien-Dindo stage 4)
  * Readmission due to a non-cardiovascular complication

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Burcharth, MD, PhD, Principal Investigator — Zealand University Hospital
Locations (1):
- Department of Surgery, Zealand University Hospital, Køge, Denmark

REFERENCES:
- [Background] Huddart S, Peden CJ, Swart M, McCormick B, Dickinson M, Mohammed MA, Quiney N; ELPQuiC Collaborator Group; ELPQuiC Collaborator Group. Use of a pathway quality improvement care bundle to reduce mortality after emergency laparotomy. Br J Surg. 2015 Jan;102(1):57-66. doi: 10.1002/bjs.9658. Epub 2014 Nov 10. PMID 25384994
- [Background] Lord JM, Midwinter MJ, Chen YF, Belli A, Brohi K, Kovacs EJ, Koenderman L, Kubes P, Lilford RJ. The systemic immune response to trauma: an overview of pathophysiology and treatment. Lancet. 2014 Oct 18;384(9952):1455-65. doi: 10.1016/S0140-6736(14)60687-5. Epub 2014 Oct 17. PMID 25390327
- [Background] Preiser JC, Ichai C, Orban JC, Groeneveld AB. Metabolic response to the stress of critical illness. Br J Anaesth. 2014 Dec;113(6):945-54. doi: 10.1093/bja/aeu187. Epub 2014 Jun 26. PMID 24970271
- [Background] Marik PE, Bellomo R. Stress hyperglycemia: an essential survival response! Crit Care Med. 2013 Jun;41(6):e93-4. doi: 10.1097/CCM.0b013e318283d124. No abstract available. PMID 23685597
- [Background] Hassan-Smith Z, Cooper MS. Overview of the endocrine response to critical illness: how to measure it and when to treat. Best Pract Res Clin Endocrinol Metab. 2011 Oct;25(5):705-17. doi: 10.1016/j.beem.2011.04.002. PMID 21925072
- [Background] Gibbison B, Angelini GD, Lightman SL. Dynamic output and control of the hypothalamic-pituitary-adrenal axis in critical illness and major surgery. Br J Anaesth. 2013 Sep;111(3):347-60. doi: 10.1093/bja/aet077. Epub 2013 May 9. PMID 23661405
- [Background] Munzel T, Sinning C, Post F, Warnholtz A, Schulz E. Pathophysiology, diagnosis and prognostic implications of endothelial dysfunction. Ann Med. 2008;40(3):180-96. doi: 10.1080/07853890701854702. PMID 18382884
- [Background] Ekeloef S, Larsen MH, Schou-Pedersen AM, Lykkesfeldt J, Rosenberg J, Gogenur I. Endothelial dysfunction in the early postoperative period after major colon cancer surgery. Br J Anaesth. 2017 Feb;118(2):200-206. doi: 10.1093/bja/aew410. PMID 28100523
- [Background] McIlroy DR, Chan MT, Wallace SK, Symons JA, Koo EG, Chu LC, Myles PS. Automated preoperative assessment of endothelial dysfunction and risk stratification for perioperative myocardial injury in patients undergoing non-cardiac surgery. Br J Anaesth. 2014 Jan;112(1):47-56. doi: 10.1093/bja/aet354. Epub 2013 Oct 29. PMID 24172055